CLINICAL TRIAL: NCT07343908
Title: An RCT: Impact of Chia Seeds on Human Breast Milk Composition
Brief Title: Impact of Chia Seeds on Human Breast Milk Composition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Presbyterian Health Foundation (Unknown); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Chia Impact
Record Dates: First submitted 2025-12-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight; Breastfeeding, Exclusive
Keywords: Obesity and Overweight; Breastfeeding, Exclusive; Breastmilk; Body Composition; Infant Growth
MeSH Terms: conditions — Obesity; Overweight; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - no intervention (No Intervention): This arm is the control arm that will not receive food-based dietary intervention
- Chia Seeds (Experimental): This group will receive the food-based intervention
  Interventions: Dietary Supplement: Chia seeds

INTERVENTIONS:
Dietary Supplement: Chia seeds — Chia seeds will be given to lactating mothers.
  Arms: Chia Seeds

SUMMARY:
The investigators' over-arching hypothesis is that mechanical and compositional properties of chia seeds supplemented during lactation diminish obesity-induced intestinal inflammation and barrier dysfunction. The investigators hypothesize these changes will result in: 1) reduced maternal systemic inflammation (serum CRP and IL-6) and increased gut microbial diversity and richness, 2) reduced HM fat and inflammatory markers, metrics the research team have demonstrated differ in tandem with maternal metabolic health and 3) improved infant growth/body composition. To test these hypotheses, investigators will evaluate chia seed supplementation during lactation in a 6wk multi-site pilot RCT (Aim 1) and through translational studies using human enteroids (Aim 2).

DETAILED DESCRIPTION:
Childhood metabolic disease has become a progressively serious global health challenge. The investigators' preliminary data reveal maternal metabolic dysfunction and poor diet are associated with increased human milk fat, proinflammatory markers, and altered microbiota, potentially contributing to transmission of metabolic susceptibility to offspring, while their studies in animal models demonstrate associations between milk composition and offspring metabolic health may be a mechanism by which lactational programming dictates offspring metabolic susceptibility. The investigators' long-term goal is to identify easy-to-implement maternal dietary interventions to optimize offspring development and prevent childhood metabolic disease. Chia seeds contain fiber, polyphenols, -3 polyunsaturated fatty acids, and bioactive peptides, and, through a multitude of mechanisms, improve the metabolic health of those with type 2 diabetes and obesity. This project will test the hypotheses that (Aim 1) 6wks of chia seed supplementation will impact obese, lactating mothers' metabolic health, milk composition, and infant growth, and (Aim 2) chia seed polyphenols and bioactive peptides will reduce permeability, inflammation, and oxidative stress, as well as ATP generating metabolism, in human enteroids, at homeostasis and during in vitro lipotoxicity. Further, investigators will utilize a luciferase-reporter assay to evaluate whether chia seed bioactives function via activation of extraoral bitter taste receptors. Successful completion of this project will inform future maternal lactational interventions that are practical and effective in reducing offspring susceptibility to childhood obesity and diabetes, supporting feasibility for a multidisciplinary, collaborative grant focused on the metabolic health of mother-infant dyads.

ELIGIBILITY:
Inclusion Criteria:

* pre-pregnancy BMI >25 kg/m²
* Maternal age 18 - 45 years at time of delivery
* Singleton pregnancy
* Vaginal delivery
* Intention to breast feed for at least three months
* No prescription medications that may interfere with gut microbiome
* Not taking antibiotics for ≥ 1 week prior to each visit
* No chia seed supplements during pregnancy

Exclusion Criteria:

* Inability to understand English
* Preterm or post-term birth (gestational age <37 or >42 weeks)
* Congenital or other defect or medical condition that would affect the mother's ability to produce milk or the infant's growth or ability to breastfeed
* Infant eating more than 12 ounces of any liquid other than breast milk in the two weeks prior to each study visit
* Taking Antibiotics (all), Proton pump inhibitors/H2 blockers, Metformin, NSAIDs, Statins, SSRIs and tricyclic antidepressants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Breast milk | 6 weeks
  Breast milk composition primarily macronutrient composition (total fat, total carbohydrate, total protein along with caloric density). Additionally, markers of inflammation (IL-6 and CRP) along with metabolic health (glucose and insulin) will be measured in milk from the collection of a complete breast expression (~1 to 2 ounces).
Breast Milk | 6 weeks
  Changes in breast milk will be investigated (both macro nutrients and small bioactive). Macronutrient composition will encompass total fat, protein and carbohydrate, along with caloric density. Small bioactives will include glucose, insulin, CRP and IL-6. This will be measured by collecting breast milk from a complete breast expression (~1 to 2 ounces).

SECONDARY OUTCOMES:
Maternal serum levels following 6 week Chia seed intervention | 6 weeks
  Baseline and 6 weeks post intervention maternal serum (~5 ml) will be collected. Maternal serum will be measured for lipids (cholesterol, triglycerides, HDL, LDL) along with markers of inflammation (IL-6 and CRP) and metabolic health (insulin and glucose).

CONTACTS AND LOCATIONS:
Overall Officials: David A Fields, Phd, Principal Investigator — University of Oklahoma; Kathy Burge, Phd, Principal Investigator — University of Oklahoma Health Sciences; Paige H Berger, Phd, RDN, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No